CLINICAL TRIAL: NCT06120998
Title: Dynamic Changes of Functional Outcome and Generic Quality of Life After Arthroscopic Rotator Cuff Repair: a Longitudinal Study.
Brief Title: Quality of Life After Arthroscopic Rotator Cuff Repair
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG8L0901
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2023-10

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tears; quality of life; ultrasound; MRI
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rotator cuff tears pending for arthroscopic rotator cuff repair: This is a Longitudinal Study. Patients were evaluated by orthopedic surgeons as having a rotator cuff tear, confirmed by magnetic resonance imaging (MRI) or ultrasound. If the patients required surgery and were willing to participate in the trial, the research assistant provided informed consent. The exclusion criteria were as follows.
  1. Acromioclavicular arthritis requiring distal clavicular resection.
  2. Severe glenohumeral arthritis (Hamada classification grade 3 or higher)15.
  3. History of shoulder fracture.
  4. Absolute contraindications to MRI, such as claustrophobia, pacemakers, neurostimulators, drug infusion pumps, artificial inner ear implants, and metallic implants.
  Interventions: Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair — All patients were placed in a semi-sitting position. Initially, a posterior portal was established to explore the inside of the joint, a lateral portal was created for the removal of subacromial bursa, and an additional anterior portal was created for repairing the tendons. Measurements were taken to determine the extent of rotator cuff damage, including its anterior-posterior and medial-lateral dimensions. In cases where complete repair was possible, a single-row or double-row repair technique was used depending on the degree of tendon damage. For situations where complete repair was not feasible, partial repair was performed. If the tendon could be stretched after relaxation, it was repaired to an anatomical position near the bone bed with the assistance of acellular dermal reinforcement. However, if the tendon lacked elasticity and was fully retracted upon relaxation, acellular dermis was used to bridge the tendon back to the anatomical position.

SUMMARY:
The goal of this longitudinal study is to understand the postoperative quality of life and dynamic trajectory of shoulder function in individuals with rotator cuff tears.

DETAILED DESCRIPTION:
Rotator cuff tears (RCTs) involve rupture of shoulder tendons or muscles, leading to pain and weakness. Its prevalence increases with age and is influenced by factors such as handedness, obesity, and smoking. Although conservative treatments are common, surgery aims to restore function. However, limited research has been conducted on postoperative psychological and social changes. Patient-reported outcome (PRO) and health-related quality of life (HRQOL) assessments are gaining importance, offering comprehensive insights into patient experiences.

This longitudinal study will include 200 randomized controlled trials (RCTs) of patients who undergo surgery. Demographics, physical examinations, and scales, such as ASES, WORC, WHOQOL-BREF, and EQ-5D, are collected preoperatively and at 2 weeks and 3, 6, 9, and 12 months postoperatively. MRI is used to assess postoperative healing at 6 months. Statistical analyses are performed using SAS software encompassing chi-square, t-tests, linear mixed effects models, and subgroup analyses to identify determinants of postoperative quality of life and functionality.

ELIGIBILITY:
Inclusion Criteria:

-Patients were evaluated by orthopedic surgeons as having a rotator cuff tear between August 2021 and July 2022, confirmed by magnetic resonance imaging (MRI) or ultrasound. If the patients required surgery and were willing to participate in the trial, the research assistant provided informed consent.

Exclusion Criteria:

1. Acromioclavicular arthritis requiring distal clavicular resection.
2. Severe glenohumeral arthritis (Hamada classification grade 3 or higher).
3. History of shoulder fracture.
4. Absolute contraindications to MRI, such as claustrophobia, pacemakers, neurostimulators, drug infusion pumps, artificial inner ear implants, and metallic implants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were evaluated by orthopedic surgeons as having a rotator cuff tear between August 2021 and July 2022, confirmed by magnetic resonance imaging (MRI) or ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Shoulder joint angles and strength were tracked preoperatively and at 3, 6, 9, and 12 months postoperatively. | 1 year
  1. Patients were seated comfortably, and a goniometer was used to measure the active range of motion (ROM) of shoulder joint angles, including internal rotation, external rotation, abduction, extension, and flexion.
  2. Patients were seated comfortably and a manual hydraulic push-pull dynamometer was used to measure the strength of internal rotation, external rotation, abduction, extension, and flexion.

SECONDARY OUTCOMES:
Questionnaire Survey | 1 year
  The following scales were administered to the patients before surgery and at 2 weeks, as well as at 3, 6, 9, and 12 months postoperatively. Owing to notable swelling and discomfort at the surgical site and joint at the 2-week postoperative mark, measurements of shoulder joint angles and strength were not advisable.
American Shoulder and Elbow Surgeons Score (ASES Score) | 1 year
  The ASES Score has been validated for use in patients with shoulder arthritis, shoulder instability, rotator cuff tears, and in those who have undergone shoulder arthroplasty. The ASES questionnaire comprises sections evaluated by physicians and self-reported by patients. The questionnaire focused on joint pain, instability, and activities of daily living. It consists of 17 questions, including one for the pain score and ten for the daily living function assessment. The final pain score was computed using an independent formula, whereas the raw functional scores were multiplied by coefficients to derive the overall functional score. The pain and functional components were then combined to yield the total ASES score, with higher scores indicating better prognosis.
Western Ontario Rotator Cuff Index(WORC) | 1 year
  The Western Ontario Rotator Cuff Index (WORC) questionnaire is primarily designed to aid in understanding the specific symptoms and functional limitations related to rotator cuff tendon pathology. It comprises 21 questions organized into five domains: Physical Symptoms, Leisure and Recreation, Work, Social, and Emotional. Each question was scored on a scale of 0 to 100, resulting in a total score ranging from 0 to 2100. Higher scores indicated a worse prognosis. However, for the purpose of comparison with other scales, the total score is subtracted by 2100 and then divided by 21 to convert it into a percentage. In this scenario, higher scores indicate a better prognosis.
Taiwan Version of the World Health Organization Quality of Life-BREF (WHOQOL-BREF) Questionnaire | 1 year
  The Taiwan version of the WHOQOL-BREF consists of 28 questions, measuring overall Quality of Life (QOL), general health status, and 26 aspects of quality of life across four main domains: Physical Health (covering the original physical and independence domains), psychological (encompassing the original psychological and spiritual/religious/personal belief domains), Social Relationships, and Environment. Higher scores indicate better prognosis.
EQ-5D Quality of Life Questionnaire for Preoperative Utility Assessment | 1 year
  The EQ-5D is a preference-based health-related quality of life measurement tool comprising five dimensions of self-classification items and a self-assessment scale for current health status ranging from 0 to 100. Each of the five dimensions has three different levels of options and various combinations correspond to different utility values. Higher utility values indicate better prognosis

OTHER OUTCOMES:
Magnetic Resonance Imaging (MRI) Follow-up | 1 year
  At 6 months postoperatively, a musculoskeletal radiologist specializing in soft tissue assessment will perform MRI to determine whether there is a re-tear of the rotator cuff, assess tendon retraction20, evaluate fat infiltration using the Goutallier classification21-23, and measure muscle atrophy24. Among these, the most crucial imaging indicator is the presence of a re-tear, which relates to the extent of postoperative functional recovery and subsequently influences changes in the psychological state. According to previous research, the optimal time for evaluating the degree of rotator cuff healing is 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Po-Cheng Chen, M.D., M.P.H., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Po-Cheng Chen, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Harris JD, Pedroza A, Jones GL; MOON (Multicenter Orthopedic Outcomes Network) Shoulder Group. Predictors of pain and function in patients with symptomatic, atraumatic full-thickness rotator cuff tears: a time-zero analysis of a prospective patient cohort enrolled in a structured physical therapy program. Am J Sports Med. 2012 Feb;40(2):359-66. doi: 10.1177/0363546511426003. Epub 2011 Nov 17. PMID 22095706
- [Result] Rhee YG, Cho NS, Yoo JH. Clinical outcome and repair integrity after rotator cuff repair in patients older than 70 years versus patients younger than 70 years. Arthroscopy. 2014 May;30(5):546-54. doi: 10.1016/j.arthro.2014.02.006. Epub 2014 Mar 14. PMID 24630958
- [Result] Chung SW, Park JS, Kim SH, Shin SH, Oh JH. Quality of life after arthroscopic rotator cuff repair: evaluation using SF-36 and an analysis of affecting clinical factors. Am J Sports Med. 2012 Mar;40(3):631-9. doi: 10.1177/0363546511430309. Epub 2011 Dec 21. PMID 22190415
- [Result] Kolk A, Wolterbeek N, Auw Yang KG, Zijl JA, Wessel RN. Predictors of disease-specific quality of life after arthroscopic rotator cuff repair. Int Orthop. 2016 Feb;40(2):323-9. doi: 10.1007/s00264-015-2996-z. Epub 2015 Oct 27. PMID 26508496